CLINICAL TRIAL: NCT00142207
Title: The Efficacy and Cost-effectiveness of Malaria Prevention in Pregnancy in an Area of Low and Unstable Transmission in Kabale, Uganda: Use of Intermittent Preventive Treatment and Insecticide-treated Nets.
Brief Title: Preventing Malaria During Pregnancy in Epidemic-prone Areas.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Ministry of Health, Uganda (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITDCVG32
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria, Falciparum
Keywords: malaria; pregnancy; intermittent preventive treatment; insecticide-treated nets
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Insecticide-Treated Bednets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Drug: Intermittent preventive treatment:sulphadoxine-pyrimethamine
  Interventions: Drug: Intermittent preventive treatment:sulphadoxine-pyrimethamine
- 2 (Active Comparator): Device: Insecticide-treated mosquito bed net
  Interventions: Device: Insecticide-treated mosquito bed net
- 3 (Active Comparator): Combination of Drug + Device:
  Drug: Intermittent preventive treatment:sulphadoxine-pyrimethamine Device: Insecticide-treated mosquito bed net
  Interventions: Drug: Intermittent preventive treatment:sulphadoxine-pyrimethamine; Device: Insecticide-treated mosquito bed net

INTERVENTIONS:
Drug: Intermittent preventive treatment:sulphadoxine-pyrimethamine — Two doses given twice during pregnancy (once in the second trimester, and once in the third trimester). Oral medication in tablet form: single daily dose given on each occasion
  Arms: 1; 3
Device: Insecticide-treated mosquito bed net — Insecticide-treated mosquito bed net
  Arms: 2; 3

SUMMARY:
The purpose of this study is to compare the efficacy and cost-effectiveness of three alternative strategies for the prevention of malaria during pregnancy in an epidemic-prone area of low transmission in the East African Highlands.

The strategies being compared are:

* intermittent preventive treatment with sulfadoxine-pyrimethamine (IPT-SP)
* an insecticide treated net (ITN), and
* intermittent preventive treatment with SP plus an ITN

In addition to the main individually-randomised trial, outcome data was subsequently also gathered on pregnant women whose houses where sprayed with indoor residual insecticides (IRS) as part of a non-randomised district-wide control programme to compare the impact of IRS with the three intervention arms.

DETAILED DESCRIPTION:
Susceptibility to malaria infection during pregnancy and the severity of clinical manifestation are determined by the level of pre-pregnancy immunity, which depends on intensity and stability of malaria transmission. Most intervention trials to prevent malaria during pregnancy have been conducted in areas of intense transmission. The results of trials conducted in high-transmission areas may not be applicable to low transmission areas, where malaria is less frequent but the risk of spontaneous abortion and stillbirth is very high in women of all parities due to lack of sufficient malaria immunity. Routine chemoprophylaxis is generally not recommended in areas of unstable malaria transmission. However, intermittent treatment with an effective anti-malarial drug may be beneficial, especially during periods of malaria transmission. Little work has been carried out amongst pregnant women living in areas of low and unstable transmission in Africa. No data are available on the cost-effectiveness of malaria control in low transmission settings.

This study will compare the efficacy and cost effectiveness of three preventive strategies for the control of malaria during pregnancy in low-transmission settings. The study is located in Kabale district, a highland area in SW Uganda.

Women attending antenatal care are randomised to receive either:

* intermittent preventive treatment with sulfadoxine-pyrimethamine (IPT-SP)
* an insecticide treated net (ITN), or
* intermittent preventive treatment with SP and an ITN. It is hypothesized that when combined with IPT-SP, the additional impact of ITNs by reducing exposure may be greatest where the intensity of transmission is low.

In addition to the main individually-randomised trial, outcome data was subsequently also gathered on pregnant women whose houses where sprayed with indoor residual insecticides (IRS) as part of a non-randomised district-wide control programme to compare the impact of IRS with the three intervention arms.

The study aims to identify the most effective intervention strategies suited to areas characterised by low and unstable transmission. Research findings should be applicable to other hypoendemic areas of the East African highlands.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women whose pregnancies are at <27 weeks gestation at first antenatal booking
* Permanent resident in study area
* Informed consent

Exclusion Criteria:

* Late presentation: pregnancies more than 26 weeks gestation at first antenatal booking
* Severe anaemia (Hb<70g/L) on enrolment
* Previous reaction to a sulfa-drug (e.g. sulphadoxine-pyrimethamine, septrin)
* History of severe skin reaction to any drug
* Current (or history) of severe disease (e.g. hepatitis, jaundice, TB, AIDS)

Withdrawal Criteria:

* Withdrawal of consent
* Women developing severe anaemia (Hb<70g/L)during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4775 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
mean birthweight | April 2004-Jan 2007
prevalence of low birthweight | April 2004 - Jan 2007

SECONDARY OUTCOMES:
maternal anaemia - mean Hb at gestational age 36 weeks, prevalence of Hb<100g/L at gestational age 36 weeks | Feb 2003 - Jan 2007
spontaneous abortions | Feb 2003 - Jan 2007
stillbirths | April 2003-Jan 2007

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Ndyomugyenyi, MBChB, PhD, Principal Investigator — Vector Control Division, Ministry of Health, Uganda; Sian E Clarke, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine, University of London, UK; Pascal Magnussen, MD, Principal Investigator — DBL - Institute for Health Research and Development, Denmark; Kristian Schultz Hansen, PhD, Principal Investigator — DBL - Institute for Health Research and Development, Denmark
Locations (1):
- Kabale District Health Services (antenatal clinics at selected sites), Kabale, Kabale District, Uganda

REFERENCES:
- [Background] Ndyomugyenyi R, Clarke S, Chandramohan D, Twesigomwe T & Magnussen P. (2005). Epidemiology of pregnancy-associated malaria in the Ugandan highlands [abstract]. Acta Tropica, Suppl 95: S448.
- [Derived] Hansen KS, Ndyomugyenyi R, Magnussen P, Clarke SE. Cost-effectiveness analysis of three health interventions to prevent malaria in pregnancy in an area of low transmission in Uganda. Int Health. 2012 Mar;4(1):38-46. doi: 10.1016/j.inhe.2011.10.001. PMID 24030879
- [Derived] Ndyomugyenyi R, Clarke SE, Hutchison CL, Hansen KS, Magnussen P. Efficacy of malaria prevention during pregnancy in an area of low and unstable transmission: an individually-randomised placebo-controlled trial using intermittent preventive treatment and insecticide-treated nets in the Kabale Highlands, southwestern Uganda. Trans R Soc Trop Med Hyg. 2011 Nov;105(11):607-16. doi: 10.1016/j.trstmh.2011.07.012. Epub 2011 Oct 2. PMID 21962292